CLINICAL TRIAL: NCT05340309
Title: A Phase II Study of Subcutaneous Atezolizumab in NSCLC Patients Using a Decentralized Clinical Trial Model
Brief Title: Subcutaneous Atezolizumab for the Treatment of Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2N-21-9; NCI-2022-02425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2N-21-9 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab and recombinant human hyaluronidase) (Experimental): Patients receive atezolizumab and recombinant human hyaluronidase SC over 3-8 minutes on day 1. Cycles repeat every 3 weeks for 1 year (early-stage lung cancer) or up to 2 years (late-stage lung cancer) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab and Recombinant Human Hyaluronidase; Other: Survey Administration

INTERVENTIONS:
Biological: Atezolizumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: Atezolizumab + rHuPH20; Atezolizumab and Hyaluronidase; Atezolizumab with rHuPH20; Atezolizumab-rHuPH20; Atezolizumab/rHuPH20 Co-formulation; Recombinant Human Hyaluronidase Mixed with Atezolizumab; Tecentriq/rHuPH20
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial tests whether subcutaneous atezolizumab can be effectively given at home with medical care provided primarily using telemedicine in patients with non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. This study may help determine if a telemedicine based approach that gives atezolizumab at home using a version of the drug designed for subcutaneous injection under the skin is safe and feasible.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of home administration by a healthcare provider (HCP) of atezolizumab and recombinant human hyaluronidase (subcutaneous atezolizumab) at a dose of 1875 mg every 3 weeks (Q3W).

II. To determine the feasibility of home administration, by mobile nursing, of subcutaneous atezolizumab at a dose of 1875 mg Q3W.

SECONDARY OBJECTIVES:

I. To determine patient satisfaction with home administration of atezolizumab. II. To determine healthcare provider and mobile nurse satisfaction with home administration of atezolizumab.

III. To determine the feasibility of a cancer clinical trial conducted under a decentralized model with telehealth assessments.

EXPLORATORY OBJECTIVES:

I. To determine the patient enrollment and retention rate for a decentralized clinical trial.

II. To determine the relationship between patient physical activity and toxicity.

III. To compare patient, infusion nurse, and pharmacist time spent in care during in office and home administration cycles.

IV. To compare efficacy of subcutaneous (SC) atezolizumab with known efficacy of intravenous (IV) atezolizumab.

OUTLINE:

Patients receive atezolizumab and recombinant human hyaluronidase SC over 3-8 minutes on day 1. Cycles repeat every 3 weeks for 1 year (early-stage lung cancer) or up to 2 years (late-stage lung cancer) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) patients who are eligible for treatment with atezolizumab for approved indications. These include the following:

  * Locally advanced or metastatic 1st line patients whose tumors have high PD-L1 expression (PD-L1 stained >= 50% of tumor cells [TC >= 50%] or PD-L1 stained tumor-infiltrating immune cells [IC] covering >= 10% of the tumor area [IC >= 10%]), as determined by an Food and Drug Administration (FDA) - approved test, with no EGFR or ALK genomic tumor aberrations
  * For the treatment of adult patients with metastatic NSCLC who have disease progression during or following platinum-containing chemotherapy. Patients with EGFR or ALK genomic tumor aberrations should have disease progression on FDA-approved therapy for NSCLC harboring these aberrations prior to receiving
  * For adjuvant treatment following resection and platinum-based chemotherapy for adult patients with stage II to IIIA NSCLC whose tumors have PD-L1 expression on >= 1% of tumor cells, as determined by an FDA-approved test
* Be willing and able to provide written informed consent/assent for the trial
* Be at least 18 years of age on day of signing informed consent
* Have detectable disease based on computed tomography (CT) and/or positron emission tomography (PET) scan
* Have ready access wifi or cellular data plan
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Ability to comply with the study protocol, in the investigator's judgment
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1500/uL) without granulocyte colony-stimulating factor support (obtained within 14 days prior to initiation of study treatment)
* Lymphocyte count >= 0.5 x 10^9/L (500/uL) (obtained within 14 days prior to initiation of study treatment)
* Platelet count >= 100 x 10^9/L (100,000/uL) without transfusion (obtained within 14 days prior to initiation of study treatment)
* Hemoglobin >= 90 g/L (9 g/dL) (obtained within 14 days prior to initiation of study treatment)

  * Patients may be transfused to meet this criterion
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) =< 2.5 x upper limit of normal (ULN) with the following exceptions (obtained within 14 days prior to initiation of study treatment):

  * Patients with documented liver metastases: AST and ALT =< 5 x ULN
  * Patients with documented liver or bone metastases: ALP =< 5 x ULN
* Serum bilirubin =< 1.5 x ULN with the following exception (obtained within 14 days prior to initiation of study treatment)

  * Patients with known Gilbert disease: serum bilirubin =< 3 x ULN
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 30 mL/min (calculated using the Cockcroft-Gault formula) (obtained within 14 days prior to initiation of study treatment)
* Serum albumin >= 25 g/L (2.5 g/dL) (obtained within 14 days prior to initiation of study treatment)
* For patients not receiving therapeutic anticoagulation: International normalized ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 x ULN (obtained within 14 days prior to initiation of study treatment)
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception

Exclusion Criteria:

* History of leptomeningeal disease
* Untreated or treatment refractory brain metastases
* Uncontrolled tumor-related pain

  * Patients requiring pain medication must be on a stable regimen at study entry
  * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  * Patients with indwelling catheters (e.g., PleurX) are allowed
* Patients with known HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/uL, and have an undetectable viral load
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than lung cancer within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival [OS] rate > 90%), such as adequately treated carcinoma in situ of the cervix or bladder, non-melanoma skin carcinoma, localized prostate or resected differentiated thyroid cancer, ductal or lobular carcinoma in situ, or stage I uterine cancer
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic IV antibiotics within 2 weeks prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Treatment with investigational therapy within 28 days prior to initiation of study treatment. However, Covid-19 vaccines administered under an FDA emergency use authorization are permitted
* Current treatment with anti-viral therapy for hepatitis B virus (HBV)
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment

  * Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment
* Intact normal skin without potentially obscuring tattoos, pigmentation, or lesions in the area for intended injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) of home administration by a healthcare provider (HCP) of subcutaneous atezolizumab | Up to 30 days after last dose
  Determined by rates of grade 3 or greater non-hematologic AE assessment by clinical assessment. Grading will be based on the NCI CTCAE v5.0 .
Successful completion of home drug administration visits within the specified window | Up to 2 years
  The number of successfully completed home visits per patient and the number of patients who successfully completed all home administrations will be calculated and reported.

SECONDARY OUTCOMES:
Patient satisfaction with home administration of atezolizumab | At end of cycle 3 and cycle 6 (each cycle is 21 days)
  Patients will be surveyed at the end of cycle 3 and cycle 6 on satisfaction with the treatment process.
Healthcare provider and mobile nurse satisfaction with home administration of atezolizumab | At end of cycle 3 and cycle 6 (each cycle is 21 days)
  Pharmacists and treating nurses will be surveyed at the end of cycle 3 and cycle 6 on time spent in drug preparation and administration as well as satisfaction with treatment administration.

OTHER OUTCOMES:
Overall response rate | Up to 2 years
  Overall response rate (confirmed partial and complete responses) will be assessed. All responses must be confirmed on subsequent scan to be considered a true response. Tumor response will be assessed using RECIST 1.1.
Progression free survival rate | Up to 2 years
  Defined as from date of start of study to the first documented disease progression according to RECIST 1.1 or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Nieva, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States